CLINICAL TRIAL: NCT03129945
Title: Comparison of Nifedipine Versus Indomethacin for Acute Preterm Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: University of California, San Francisco (Other); University of California, Davis (Other); University of California, San Diego (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Judith H Chung, MD, Professor, Division of Maternal Fetal Medicine, Dept OBGYN, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1085; UC Reliance 857 (Other: University of California)
Record Dates: First submitted 2015-01-05; First posted 2017-04-26 (Actual); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Obstetric Labor, Premature
Keywords: Obstetric Labor, Premature; Tocolytic Agents
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Nifedipine; Indomethacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nifedipine (Active Comparator): Participants will be given this medication orally
  Interventions: Drug: Nifedipine
- Indomethacin (Active Comparator): Participants will be given this medication orally
  Interventions: Drug: Indomethacin

INTERVENTIONS:
Drug: Nifedipine — Subjects will be given nifedipine 10mg orally and repeated every 20 minutes for a maximum dose of 30mg in the first hour followed by 20mg every 6 hours for the first 48 hours.
  Other Names: Procardia
  Arms: Nifedipine
Drug: Indomethacin — Those randomized to indomethacin will be given 100mg orally as a loading dose followed by 50mg every 6 hours for the first 48 hours of treatment.
  Other Names: Indocin
  Arms: Indomethacin

SUMMARY:
The purpose of this research study is to determine the best medication to stop preterm labor. Recent studies have identify nifedipine and indomethacin as the two medications that are most likely to delay delivery for 48 hours, decrease maternal side effects and decrease some complications related to preterm delivery to the neonate. Both of these medications are commonly used to stop pre-term labor, therefore it has become our institution's standard to use these two medications in the setting of preterm labor. There have been limited studies comparing these two medications directly.

A total of 450 participants will be asked to participate across all study sites.

DETAILED DESCRIPTION:
There are about 10 million births that occur before 37 weeks (prior to full term gestation) that occur annually worldwide. More than 1 million infants die from complications related to preterm birth. Tocolytics, medications that stop preterm labor, have been well studied. Results regarding prolongation of pregnancy are varied, but tocolytics have been shown to delay delivery for 48 hours, allowing time to administer corticosteroids. ACOG (American Congress of Obstetrics and Gynecologists) recommends giving tocolytics to provide time for corticosteroid administration, transfer to tertiary level care and to allow for magnesium infusion to protect the neonatal brain. Corticosteroid administration when the course is completed (48 hours from first dose) decreases some of the major risks associated with prematurity.

Recent meta-analyses have shown of the commonly used tocolytics, calcium channel blockers and prostaglandin inhibitors ranked consistently among the top three medications in several categories including delaying delivery by 48 hours. There have been only two published randomized control studies to date that have directly compared these two tocolytics. These studies lacked power and standardization to provide clinical guidelines. There is a high neonatal mortality and morbidity along with exceedingly high hospital costs associated with complications related to preterm birth, so it is important to intervene with superior medications. Here the investigators propose a multi institutional (based within the University of California system) randomized controlled study to directly compare nifedipine (most commonly used calcium channel blocker) to indomethacin (most commonly used prostaglandin inhibitor).

Objective:

The Investigator's objective is to compare the prolongation of pregnancy by 48 hours after women are diagnosed with preterm labor prior to 32 weeks gestational age and treated with either nifedipine or indomethacin. Investigators hypothesize that indomethacin will significantly arrest preterm labor by 48 hours in more women compared to nifedipine. The primary outcomes measures will be delaying preterm delivery by 48 hours; secondary outcomes measures will include delay of delivery by 7 days and decreasing delivery before 37 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy. A twin pregnancy reduced to singleton (either spontaneously or therapeutically) before 140 weeks by gestational age (see dating below) is acceptable.
* Gestational age at randomization between 240 weeks to 315 weeks by using the dating determinations as below
* Preterm labor with intact membranes. Preterm labor is defined as at least 6 regular uterine contractions in 60 minutes either seen on tocodynamometer, palpated by health providers and/or subjectively felt by the patient and at least one of the following:

  1. Associated with cervical change by cervical dilation greater than or equal to 1cm OR effacement greater than or equal to 25 to 50%
  2. Cervix greater than or equal to 2cm dilated on initial digital exam
  3. At least 75% effaced on initial digital exam
  4. Short cervical length (defined by each institution's policy) as obtained by transvaginal cervical sonography [in general, this is defined as a measurement of 2.0 - 2.5 cm or less] and/or a positive fetal fibronectin test (defined as a level greater than 50ng/mL).
* Intact membranes
* 18 years of age or older

Exclusion Criteria:

* Fetal demise, or known major fetal anomaly, including cardiac anomaly and hydrops
* Maternal contraindication to nifedipine: preload cardiac lesions or maternal hypotension (systolic blood pressure less than 100 or diastolic blood pressure less than 60). A delayed dose can be given if blood pressure improves - it will be documented if dose is delayed, how long from scheduled dose it was delayed and reason for delay.
* Maternal contraindication to indomethacin: platelet dysfunction or bleeding disorders, hepatic dysfunction, gastrointestinal ulcerative disease, renal dysfunction and asthma
* Obstetrical contraindication to tocolysis not already mentioned: non reassuring fetal status, severe preeclampsia or eclampsia, maternal bleeding with hemodynamic instability, chorioamnionitis, preterm premature rupture of membranes
* Participation in another interventional study that influences neonatal morbidity or mortality
* Participation in this trial earlier in the pregnancy
* Maternal allergy to either indomethacin or nifedipine
* Maternal allergy to aspirin and other NSAIDs.
* Maternal hypertension requiring treatment.
* Maternal kidney disorder that would require adjustment in magnesium dosing.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Wing, MD, Principal Investigator — University of California, Irvine; Mary Norton, MD, Principal Investigator — University of California, San Francisco; Gladys (Sandy) Ramos, MD, Principal Investigator — University of California, San Diego; Aisling Murphy, MD, Principal Investigator — University of California, Los Angeles; Veronique Tache, MD, Principal Investigator — University of California, Davis
Locations (5):
- United States (5):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Irvine, Orange, California
  - University of California, Davis, Sacramento, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from January 17, 2017, to February 24, 2018.
Period: Overall Study
Arm/Group | Nifedipine | Indomethacin
Started | 15 | 21
Completed | 15 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nifedipine | Indomethacin | Total
Number analyzed (Participants) | 15 | 21 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 21 | 36
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 21 | 36
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 21 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Delay of Preterm Delivery by 48 Hours.
Description: 1. To compare the prolongation of pregnancy by 48 hours after women are diagnosed with threatened preterm labor prior to 32 weeks gestational age and treated with either nifedipine or indomethacin. The primary outcome measured will be delay of (preterm delivery) by 48 hours.
Time Frame: Participants will be followed for the duration of the hospital stay, an expected average of 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Nifedipine | Indomethacin
Number analyzed (Participants) | 15 | 21
Participants | 15 | 21

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through study completion, for an average of 1 week.
Description: Adverse event definition did not differ from the clinicaltrials.gov definitions.
Arm/Group | Nifedipine | Indomethacin
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/21
Other Adverse Events (participants affected / at risk) | 1/15 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nifedipine (N=15) | Indomethacin (N=21)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT03129945/Prot_SAP_000.pdf